CLINICAL TRIAL: NCT04883775
Title: 89Zr-DFO-HuMab-5B1 (MVT-2163) Imaging in Pancreatic Cancer or Other CA19-9 Positive Malignancies
Brief Title: Study of a New Technique for Imaging Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-342
Record Dates: First submitted 2021-05-10; First posted 2021-05-12 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer; Tumors That Express CA19-9
Keywords: 89Zr-DFO-HuMab-5B1 (MVT-2163); Imaging; MVT-5873; 20-342
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a phase I, open label, nonrandomized, dose-escalation trial of a fixed dose of MVT-2163 (89Zr-DFO-HuMab-5B1) and varying antibody masses of MVT-5873 (HuMab-5B1), designed to identify an optimal dose (total antibody mass) and optimal timing, for tumor imaging. This trial will include dose escalation, which includes up to 5 cohorts, an expansion phase, a re-entry phase, and a pre-surgery phase.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 89Zr-DFO-HuMab-5B1 (MVT-2163) Imaging (Experimental): All subjects will receive a single, fixed, intravenous dose of MVT-2163, consisting of 3 mg (nominal mass - actual mass administered will likely vary between 2.0 and 2.5 mg) of MVT-2163 radiolabeled from 5 mCi to no less than 1.0 mCi (adjusted as of 16-Mar 2017) of 89Zr.Cohort 1 subjects will receive MVT-2163, with no MVT-5873 pre-dosing. Subjects in subsequent cohorts 2 and 3 will receive a dose of MVT-5873 15 minutes, ~ 2 hours, and ~4 hours prior to administration of MVT-2163. Future cohorts 4 and 5 may evaluate alternate time frames. Other cohorts may evaluate administration of MVT-5873 one week prior (D-7) to the day of MVT-2163 administration and a second administration of MVT-5873 the day of (D0) MVT-2163 administration. The re-entry (RE) and pre-surgery (PS) cohorts will administer MVT-2163 3 ± 1 hour after administration of MVT-5873.
  Interventions: Drug: MVT-2163; Drug: MVT-5873

INTERVENTIONS:
Drug: MVT-2163 — MVT-2163 is administered intravenously as a PET imaging agent.
  Other Names: 89Zr-DFO-HuMab-5B1
Drug: MVT-5873 — MVT-5873 will be administered intravenously over at least 60 minutes.

SUMMARY:
The purpose of this study is to see how well the experimental imaging agent 89Zr-DFO-HuMab-5B1 attaches to pancreatic tumors, and to find out whether PET/CT scans done with this imaging agent produce better images of cancer.

ELIGIBILITY:
Inclusion Criteria:

PART I : ESCALATION, EXPANSION, RE-ENTRY COHORTS:

* Histologically confirmed, locally-advanced, or metastatic pancreatic ductal adenocarcinoma (PDAC) or other malignancies known to express CA19-9 positive malignancies

PART II: PRE-SURGERY COHORT ONLY:

* Patients with biopsy-proven or high suspicion on imaging for pancreatic ductal adenocarcinoma (PDAC) (Stage T2 and T3)
* Patients scheduled referred to surgery or biopsy as standard of care for their pancreatic adenocarcinoma OR
* Patients with Intraductal papillary mucinous neoplasm (IPMN) referred to surgery or biopsy as standard of care.

The suspicion for pancreatic carcinoma and decision for surgery or biopsy will be based on review of imaging and clinical findings in the disease management team discussion including surgeon and radiologist.

PART I and II:

* Signed, informed consent
* Age 18 or more years
* At least one lesion by CT or MRI ≥ 2 cm, unless determine otherwise for pre-surgery cohort subjects
* CA19-9 serum level:

  * For Part I: >ULN or CA19-9 positive biopsy (optional);
  * For Part II ( presurgical cohort): CA19-9 serum level (normal or high levels are allowed) or CA19-9 positive biopsy (optional)
* ECOG performance status of 0 to 2
* Adequate laboratory parameters including:

  * Absolute neutrophil count (ANC) ≥1.5 x 10^9/L
  * Hemoglobin ≥ 9.0 g/dL (in the absence of red blood cell transfusions in the prior 14 days)
  * Platelet count >75,000/ mm^3
  * AST/SGOT, ALT/SGPT ≤2.5 x ULN, unless liver metastases are clearly present, then ≤5.0 x ULN
  * Total bilirubin ≤1.5x the upper limit of normal unless considered due to Gilbert's syndrome in which case, ≤3x the upper limit of normal
  * Creatinine (serum or plasma) ≤ 1.5 x ULN or eGFR>50 mL/min

PART I: ESCALATION, EXPANSION, RE-ENTRY COHORTS:

* Willingness to participate in collection of pharmacokinetic samples

Exclusion Criteria:

* Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Major surgery other than diagnostic surgery within 4 weeks of Study Day 1
* History of anaphylactic reaction to human, or humanized, antibody
* Other on-going cancer therapy or investigational agents (except MVT-5873)
* Known history of HIV
* Pregnant or currently breast-feeding
* Psychiatric illness/social situations that would interfere with compliance with study requirements
* Prior entry onto this protocol 3 or more times (e.g., subjects may enter this protocol and be imaged up to 3 times)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-related adverse events as assessed | 1 year
  assessed by CTCAE v4.0
Biodistribution of MVT-2163 | 1 year
  will be determined by measuring radiation exposure for key organs and tissues

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Pandit-Taskar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only ), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

DOCUMENTS (1):
  • Informed Consent Form (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT04883775/ICF_000.pdf